CLINICAL TRIAL: NCT07081386
Title: LAPARO Analytic vs. Classic Box Trainer: A Randomized Trial on Appendicectomy Laparoscopic Skills Training
Brief Title: LAPARO Analytic vs. Classic Box Trainer on Laparoscopic Skills Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UPorto-LAPTRAIN-NSG
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Laparoscopic Surgical Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic Box Trainer Group (Other): Participants in this group will receive a single, 3-hour in-person laparoscopic training session using a Classic Box Trainer. Training will be supervised by an experienced General Surgery tutor and focused on key technical skills required for laparoscopic appendicectomy.
  Interventions: Other: Laparoscopic Training using a classic Box Trainer
- LAPARO Analytic Group (Experimental): Participants in this group will undergo a 3-hour in-person laparoscopic training session using the LAPARO Analytic simulator. The session will be supervised by an experienced General Surgery tutor and will include real-time performance analytics to guide skill acquisition relevant to laparoscopic appendicectomy.
  Interventions: Other: Laparoscopic Training using the LAPARO Analytic simulator

INTERVENTIONS:
Other: Laparoscopic Training using the LAPARO Analytic simulator — Participants in the experimental group will undergo a 3-hour in-person laparoscopic training session using the LAPARO Analytic simulator. The session will be supervised by an experienced General Surgery tutor and will include real-time performance analytics to guide skill acquisition relevant to laparoscopic appendicectomy.
  Arms: LAPARO Analytic Group
Other: Laparoscopic Training using a classic Box Trainer — Participants will receive a single, 3-hour in-person laparoscopic training session using a Classic Box Trainer. Training will be supervised by an experienced General Surgery tutor and focused on key technical skills required for laparoscopic appendicectomy.
  Arms: Classic Box Trainer Group

SUMMARY:
This randomized controlled trial investigates the effectiveness of two laparoscopic training modalities - Classic Box Trainers and the LAPARO Analytic - in teaching fundamental surgical skills for laparoscopic appendicectomy. A total of 60 first-year medical residents (interns) from Centro Hospitalar Universitário de São João (CHUSJ) will be recruited and randomly assigned to one of two training groups. One group will undergo a 3-hour in-person training session using Classic Box Trainers, while the other group will train using the LAPARO Analytic simulator, both under the supervision of experienced General Surgery tutors. The study aims to evaluate technical skill acquisition, retention, and participant satisfaction. Outcomes will be assessed through objective performance metrics and participant feedback, contributing to the optimization of laparoscopic education methods.

DETAILED DESCRIPTION:
Minimally invasive techniques have become the standard of care in elective abdominal surgery, leading to a significant increase in laparoscopic procedures. This shift presents a major training challenge, as the acquisition of core laparoscopic skills - such as hand-eye coordination via video and depth perception - requires a steep and lengthy learning curve that may be unsafe and inefficient if conducted exclusively in the operating room.

To address these limitations, simulation-based training has emerged as an effective alternative. Classic Box Trainers are widely used in surgical education, allowing for repeated, structured practice in a safe, non-clinical environment. However, recent advancements have introduced modern systems like the LAPARO Analytic, which provides real-time instrument tracking, objective scoring, and performance analytics.

Despite their growing use, there is a lack of direct comparative evidence on the training efficacy of these two modalities, particularly for initial surgical procedures such as laparoscopic appendicectomy. This randomized prospective trial aims to fill this gap by evaluating the relative effectiveness of the LAPARO Analytic versus Classic Box Trainers in the acquisition and retention of essential laparoscopic skills.

A total of 60 first-year medical residents (interns) at Centro Hospitalar Universitário de São João (CHUSJ) will be recruited via convenience sampling and voluntary sign-up. Participants will be randomly assigned using an online tool (Research Randomizer) into two groups:

Control Group (n = 30): Will receive a 3-hour in-person training session using Classic Box Trainers, supervised by an experienced General Surgery tutor.

Intervention Group (n = 30): Will receive a 3-hour in-person training session using the LAPARO Analytic simulator, also supervised by a qualified General Surgery tutor.

Participants with any previous exposure to laparoscopic surgical techniques will be excluded, as well as those who acquire such experience between recruitment and training.

The primary outcome is the quality of technical skill execution and its retention, measured using objective assessment tools. Secondary outcomes include participant satisfaction, captured via structured questionnaires. The study aims to contribute valuable evidence to inform laparoscopic training programs and guide the integration of advanced simulation technologies into surgical education.

ELIGIBILITY:
Inclusion Criteria:

* First-year medical residents (internos de ano comum) currently enrolled at Centro Hospitalar Universitário de São João (CHUSJ).
* Voluntary participation confirmed by completion of an informed consent and online registration form.
* Availability to participate in both the initial training session and the follow-up cadaveric assessment 15 days later.

Exclusion Criteria:

* Any prior exposure to laparoscopic surgical techniques formal training.
* Engagement in any laparoscopic training activities between the recruitment date and the practical evaluation session.
* Inability to attend either the scheduled training or the cadaveric assessment session.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Technical Performance Score on Laparoscopic Appendicectomy Skills using de GOALS scale | 15 days after training session
  Participants' technical skills will be assessed 15 days after training during a laparoscopic appendicectomy performed on a human cadaver. Procedures will be video-recorded and evaluated by blinded expert raters using the Global Operative Assessment of Laparoscopic Skills (GOALS) scale. Domains assessed include depth perception, bimanual dexterity, efficiency, tissue handling, and autonomy. Scores will be compared between the two groups.

SECONDARY OUTCOMES:
Procedure Completion Time | 15 days after training session
  The duration of the laparoscopic appendicectomy performed on the cadaver model will be measured in minutes and seconds. The total time required to complete the surgical task will be compared between groups to assess efficiency.
Self-Perceived Competence in Laparoscopic Skills | Immediately after cadaver procedure (Day 15)
  Participants will complete a post-training Likert-scale questionnaire assessing their self-perceived competence in performing key laparoscopic tasks: identifying the appendix, lysis of adhesions, vascular control, stump division, and safe extraction. Responses range from 1 (strongly disagree) to 5 (strongly agree).

IPD SHARING:
Plan to Share IPD: No